CLINICAL TRIAL: NCT01817868
Title: Evaluation of Efficacy, Safety and Costs of Recombinant FVIII Products Applied to Severe Hemophilia A Patients: Observational Data Collection Study Evaluating On-demand Treatment and Secondary Prophylaxis
Brief Title: Comparison of Efficacy, Safety and Costs of Recombinant FVIII Products Between On-demand and Secondary Prophylaxis Groups in Haemophilia A Patients
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16368; KG1210TR (Other: Company Internal)
Record Dates: First submitted 2013-03-12; First posted 2013-03-26 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Hemophilia
Keywords: Hemophilia; Turkey; Observational; Adult
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: Recombinant Factor VIII (Kogenate, BAY14-2222)

INTERVENTIONS:
Other: Recombinant Factor VIII (Kogenate, BAY14-2222) — All dosage, frequency and duration for drugs will be under the decision of the treating physician.

SUMMARY:
The project is an observational, multi-central, prospective, non-interventional and open-label data collection study on secondary prophylaxis with recombinant FVIII products in adolescents and adults with severe hemophilia A (FVIII < 1%).

It will be a controlled observation of patients on secondary prophylaxis versus on-demand treatment regimen. Patients will be enrolled preferably on a 1:1 basis with regards to prophylaxis and on-demand treatment.

The patient enrollment period will be 2 years with a follow-up (observation period) of 2 years for each patient. Based on the primary effectiveness parameters (joint bleeds and overall bleeds per year) an observation period of 2 years is considered sufficient although it has to be admitted that it is rather short to assess the progression of orthopedic status. Previously treated prophylaxis patients with at least 50 exposure days and patients with continuing prophylaxis treatment will be included.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severe hemophilia A (FVIII<1%) diagnosis
* Prior treatment or ongoing treatment with on-demand or prophylaxis regimens according to Turkish guidelines and requirements
* Previously treated patients with at least >50 exposure days
* Written informed consent signed by patient/legal representative

Exclusion Criteria:

* Currently on immune tolerance treatment
* Platelet count < 75,000/mm3
* Participation in another study
* Existence of inhibitors in the past and in the last currently available blood sample prior to study start (Bethesda titer < 0.6 BU/ml)
* Existence of inhibitor history in family members who also are diagnosed with hemophilia A
* Having been on primary prophylaxis as defined in the introduction
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult haemophilia patients already on treatment with commercially available recombinant FVIII products.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2013-01-04 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Median ±SD, range of number of joint bleeds per year of prophylaxis versus on-demand group | After 4 years
Mean ±SD, range of number of joint bleeds per year of prophylaxis versus on-demand group | After 4 years

SECONDARY OUTCOMES:
Number of overall bleeding episodes | After 4 years
Musculoskeletal evaluation recommended by World Federation of Hemophilia: Orthopedic Joint Score (Gilbert Score) | After 4 years
Musculoskeletal evaluation recommended by World Federation of Hemophilia: Radiological evaluation (Pettersson Score) | After 4 years
Cost-effectiveness (cost of additional joint bleed) | After 4 years
Cost-utility | After 4 years
  The costs of care of subjects with haemophilia will be evaluated adopting the perspective of the payer, i.e. the Social Security Institution [SSI].
Comparison of patient compliance between prophylaxis and on-demand therapy groups | After 4 years
Number of spontaneous bleeds | After 4 years
Quality of life as measured with the SF-36 | Baseline and after 4 years
Quality of life as measured with Hemo-QoL | Baseline and after 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.